CLINICAL TRIAL: NCT05792163
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single and Multiple Ascending Dose Study to Investigate the Safety, Tolerability, and Pharmacokinetics of SNP318 in Healthy Adult Participants
Brief Title: A First Time in Human Study of SNP318 as a Treatment for Neurodegenerative Diseases Including Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SciNeuro (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: SNP318-101
Record Dates: First submitted 2023-02-28; First posted 2023-03-31 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Neurodegenerative Diseases; Alzheimer's Disease
MeSH Terms: conditions — Neurodegenerative Diseases; Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (SNP318) (Experimental): Drug: SNP318, Dose level: Start from 1mg for single ascending dose and from 30mg for multiple ascending dose. Dose levels can be adjusted based on emerging safety, tolerability, pharmacokinetics data of previous cohorts.
  Dosage form: Capsule Route of administration: Oral
  Interventions: Drug: SNP318 (A)
- B (Placebo) (Placebo Comparator): Placebo comparator taken by participants randomized to the placebo arm in each cohort in Part 1 and Part 2.
  Interventions: Drug: Placebo (B)

INTERVENTIONS:
Drug: SNP318 (A) — Capsule for oral administration
  Arms: A (SNP318)
Drug: Placebo (B) — Placebo capsules matching the SNP318 capsules
  Arms: B (Placebo)

SUMMARY:
SNP318 is developed to treat neurodegenerative diseases including Alzheimer's disease. In the current phase 1 study, the IP is tested in healthy volunteers, and the purpose is to investigate the safety, tolerability, and PK of single and multiple ascending oral doses of SNP318.

DETAILED DESCRIPTION:
A total of approximately 86 healthy male and female adult participants aged 18 years and older will be enrolled in this study, that will be conducted in 2 parts:

Part 1-Single Ascending Dose (SAD) and Part 2 -Multiple Ascending Dose (MAD). Part 1 is subdivided into Part 1a and Part 1b. Part 1b is a cohort for cerebrospinal fluid sampling.

There are 6 cohorts planned for Part 1a SAD, 1 cohort for Part 1b SAD and 3 cohorts for Part 2 MAD.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be ≥18 years of age, at the time of signing the informed consent.
2. Participants who are overtly healthy, in the opinion of the Investigator, as determined by medical evaluation including medical history, physical examination, vital signs, ECGs and laboratory tests. Participants who do not qualify based on a reversible condition or mild intercurrent illness may be re-screened after the underlying condition is resolved.
3. Body weight between 50.0 and 120.0 kg, inclusive, if male; and between 40.0 and 120.0 kg, inclusive, if female. Body Mass Index within the range ≥19 and ≤30 kg/m2 (inclusive), at screening.
4. Female participants who engage in heterosexual intercourse must be of non-childbearing potential, defined as either surgically sterile (ie, hysterectomy, bilateral salpingectomy, or bilateral oophorectomy), OR be postmenopausal with at least 1 year of amenorrhea, OR must be using an established form of highly effective method of contraception from the time of screening until at least 90 days after the last dose of study intervention. Female participants must not be lactating and must agree to have no egg donation plan during the study and for 90 days after the last dose of study intervention.
5. Male participants must agree to use a condom when sexually active with a female partner of childbearing potential from screening until at least 90 days after the last dose of study intervention (or be surgically sterile [ie, vasectomy with documentation]; or remain abstinent, when this is in line with the preferred and usual lifestyle). Male participants should also agree not to donate sperm for the duration of the study and until at least 90 days after the last dose of study intervention.
6. Must be capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

1. Known hypersensitivity, allergy, intolerance, or idiosyncratic reaction to the study intervention, or any of the excipients contained in the intervention formulation. If any history of anaphylaxis or reaction to other agents, discussion with (and approval by) the Investigator and Sponsor is required.
2. Any concomitant disease, condition, or treatment that could interfere with the conduct of the study or that would, in the opinion of the Investigator or Sponsor, pose an unacceptable risk to the participant in the study or interfere with the interpretation of study data.
3. History of dysphagia or any gastrointestinal disease (including Gilbert's syndrome) that affects the participants ability to swallow and/or affects drug absorption.
4. Positive severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) test at any time prior to administration of the study intervention if SARS-CoV-2 test is performed.
5. Any clinically significant (at the discretion of the Investigator) abnormalities in laboratory test results. Total bilirubin value up to 1.5 times the upper normal limit of normal can be acceptable if associated with normal conjugated bilirubin value (unless the participant has documented Gilbert's Syndrome).
6. History of immunological disorders, auto-immune disorders, acquired or congenital immune deficiency, including autoimmune rheumatic disease.

   Note: participants with mild asthma controlled with occasional rescue inhaler only (no chronic therapy; no inhaled corticosteroids), and mild atopic dermatitis controlled with topic emollients only (no topical corticosteroids) are not excluded.
7. Immunization with any live vaccine within 28 days prior to administration of study intervention; or expected to require any live vaccines during study period.
8. Evidence at the initial screening visit of active or prior hepatitis B infection based on serological tests for hepatitis B surface antigen (HbsAg).
9. Positive serological tests for human immunodeficiency virus (HIV) antibody and/or hepatitis C virus (HCV) antibody at the initial screening visit.
10. Blood donation of >400 mL within 3 months before screening or >200 mL within 4 weeks before screening or plan to donate blood during study period.
11. Acute or febrile illness within 7 days prior to the first dose of study intervention or participants with evidence of active infection.
12. Evidence of an active or suspected cancer or a history of malignancy within the previous 3 years, except for the following, which did not require systemic therapy and are considered cured: nonmelanoma skin cancer, curatively treated localized prostate cancer, or other in situ cancer.
13. History of drug abuse or a positive drug abuse test result at screening or D-1.
14. History of alcohol abuse or a positive alcohol test result at screening or D-1.
15. Use of prescription medications or herbal remedies within 14 days or 5 elimination half-lives (whichever is longer) of study intervention administration or use of over the counter (OTC) drugs within 7 days of study intervention administration (apart from recommended doses of vitamin/mineral supplements, OTC analgesics, or other agents that have been discussed with and approved by the Investigator and Sponsor). Participants who used recommended doses of paracetamol/ibuprofen for acute conditions (e.g., headache) will not be excluded. Participants who have been on hormone replacement therapy (HRT) or oral contraception for a period of at least 2 months prior to the start of screening will not be excluded from the study, provided the contraceptive or HRT regimen will remain unchanged during the conduct of the study.
16. Use of any known liver enzyme inducer or liver enzyme inhibiting food or beverage (such as all citrus fruits including tangerine, grapefruit, sweet orange, lime, kumquat, citron, orange, lemon, etc., and fruit juices) within 7 days prior to administration.
17. Any major surgery within 6 months before screening, or plan to have a surgery during the study period.
18. Any other conditions that the Investigator considers may affect the participants' informed consent or adherence to the study protocol, completion of the test according to the study procedure, or the participants' participation in the test may affect the test results or their own safety.
19. Receipt of another study intervention within 1 month or 5 elimination half-lives (whichever is longer) prior to administration of the study intervention.
20. Abnormal cardiac conditions and ECG:

    i. The Fridericia algorithm corrected QT interval (QTcF) of ECG during screening period is >450 ms for males and >470 ms for females or is considered abnormal with clinical significance as determined by the Investigator.

    ii. Sustained (ie, 3 independent measurements within 30 minutes) HR (pulse) >100 or <40 bpm.

    iii. Personal and/or family history of congenital long QT syndrome or sudden cardiac death.
21. Pregnant (positive blood or urine pregnancy test at the initial screening visit or D-1).
22. Is or has an immediate family member (e.g., spouse, parent/legal guardian, sibling, or child) who is investigational site or Sponsor staff directly involved with this study.
23. Unwilling to abstain from smoking or vaping and the consumption of any caffeine or alcohol-containing food or drinks that may influence the drug metabolism from 72 hours before administration to discharge.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2023-11-29 (Actual); Study Completion 2023-11-29 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of SNP318 in healthy adult participants. Assessed by adverse events | Up to 20 days

SECONDARY OUTCOMES:
Plasma PK parameters of SNP318 in healthy adult participants. Assessed by Maximum concentration (Cmax) | Up to 20 days
Plasma PK parameters of SNP318 in healthy adult participants. Assessed by Time of maximum concentration observed (Tmax) | Up to 20 days
Plasma PK parameters of SNP318 in healthy adult participants. Assessed by Area under the concentration-time curve from time 0 to the time of the last quantifiable concentration (AUC) | Up to 20 days
Plasma PK parameters of SNP318 in healthy adult participants. Assessed by Apparent oral clearance (CL/F) | Up to 20 days
Plasma PK parameters of SNP318 in healthy adult participants. Assessed by Apparent volume of distribution at steady state (Vss/F) | Up to 20 days
Plasma PK parameters of SNP318 in healthy adult participants. Assessed by Apparent terminal phase half-life (T1/2z) | Up to 20 days
The concentration of SNP318 in CSF samples in healthy adult participants | Up to 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- CMAX Clinical Research, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No